CLINICAL TRIAL: NCT05347576
Title: A Randomized, Open-label, Single Dose, Crossover Study to Evaluate the Pharmacokinetic Profiles and Safety of CKD-393(2) in Healthy Volunteers Under Fed Conditions
Brief Title: A Study to Evaluate the Pharmacokinetic Profiles and Safety of CKD-393(2) in Healthy Volunteers Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A98_07BE2201
Record Dates: First submitted 2022-04-21; First posted 2022-04-26 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Type2Diabetes
MeSH Terms: interventions — lobeglitazone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sequence 1 (Experimental): Period 1- A single dose of 4 tablets(CKD-501 1T, D759 1T, D150 1T, D029 1T) under fed condition Period 2- A single dose of 2 tablets(CKD-393(2) 2T) under fed condition
  Interventions: Drug: CKD-393(2); Drug: CKD-501, D759, D150, D029
- sequence 2 (Experimental): Period 1- A single dose of 2 tablets(CKD-393(2) 2T) under fed condition Period 2- A single dose of 4 tablets(CKD-501 1T, D759 1T, D150 1T, D029 1T) under fed condition
  Interventions: Drug: CKD-393(2); Drug: CKD-501, D759, D150, D029

INTERVENTIONS:
Drug: CKD-393(2) — QD, PO
Drug: CKD-501, D759, D150, D029 — QD, PO

SUMMARY:
A Study to Evaluate the Pharmacokinetic Profiles and Safety of CKD-393(2) in Healthy Volunteers Under Fed Conditions

DETAILED DESCRIPTION:
A randomized, open-label, single dose, crossover study to evaluate the pharmacokinetic profiles and safety of CKD-393(2) in healthy volunteers under fed conditions

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult volunteers aged 19 ≤ ~ < 55-year-old.
2. Weight ≥55kg (man) or 45kg (woman), with calculated body mass index(BMI) of 17.5 ≤ ~ < 30.5 kg/m2.
3. Those who have no congenital diseases or chronic diseases within 3 years and have no abnormal symptoms or findings.
4. Those who are eligible for clinical trials based on laboratory(hematology, blood chemistry, serology, urology) and 12-lead ECG results at screening.

Exclusion Criteria:

1. Those who have clinically significant disease or medical history of heart failure, Hepatopathy, Type 1 Diabetes, Diabetic ketoacidosis, Edema, Renal dysfunction, galactose intolerance, glucose-galactose malabsorption. And Those who receive intravenous administration of radioactive iodine contrast agents (for intravenous urography, venous cholangiography, angiography, computed tomography using contrast agents, etc.) during clinical trial.
2. Those who have past medical history of gastrointestinal disorder (Crohn's disease, ulcerative colitis, etc. except simple appendectomy or hernia surgery), which affect the absorption of investigational drug.
3. Those who are pregnant or breastfeeding.
4. Those who are deemed inappropriate to participate in clinical trial by investigators.

Ages: 19 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2022-04-21 (Actual); Primary Completion 2022-05-02 (Actual); Study Completion 2022-05-09 (Actual)

PRIMARY OUTCOMES:
AUCt | Pre-dose(0 h), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48 (h ) hours
  Area under the concentration-time curve from time zero to time
Cmax | Pre-dose(0 h), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48 (h ) hours
  Maximum plasma concentration of the drug

CONTACTS AND LOCATIONS:
Overall Officials: Min Gul Kim, M.D, Ph.D., Principal Investigator — Chonbuk National University Hospital
Locations (1):
- Chonbuk National University Hospital, Jeonju, South Korea